CLINICAL TRIAL: NCT05158816
Title: Extracorporal Membrane Oxygenation for Critically Ill Patients With COVID-19: a Single Centre Analysis
Brief Title: Extracorporal Membrane Oxygenation for Critically Ill Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Principal Investigator, Jessa Hospital
Other Study IDs: f/2021/097
Record Dates: First submitted 2021-12-10; First posted 2021-12-15 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
Keywords: ECMO
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 patients: COVID-19 patients admitted to the ICU
  Interventions: Procedure: ECMO

INTERVENTIONS:
Procedure: ECMO — Patients undergoing extracorporeal membrane oxygenation

SUMMARY:
Retrospective single center analyses of COVID-19 patients admitted to the ICU between 01/02/2020 and 31/07/2021.

DETAILED DESCRIPTION:
All adults (>18 years) with acute hypoxaemic respiratory failure due to diagnosed COVID-19 pneumonia and admitted to ICU from 01/02/2020 until 31/07/2021 were included in the study. Following the World Health Organisation (WHO) protocol 19, laboratory confirmation of COVID-19 infection was defined as a positive result on polymerase chain reaction (PCR) assays of nasopharyngeal swab samples or bronchoalveolar lavage. Only laboratory-confirmed patients were included in the analysis.

Additional data collection

Additional collected parameters are listed below and are collected as a standard-of-care in our hospital:

* Demographics: i.e age, gender, BMI
* DNR code
* Comorbidities: smoking, obesity, hypertension, diabetes, cardiovascular disease, respiratory disease, malignancies, renal failure (AKI), liver failure, gastrointestinal disease, neurological conditions, mental state, other
* Symptoms at the time of admission to ICU: i.e fever, body temperature, dyspnoea, headache, diarrhea etc…
* Laboratory results of all standard parameters measured
* Treatment: antiviral agents, antibiotics, etc…
* Complications: shock, heart failure, sepsis, stroke, etc…
* Ventilation: method, PEEP, FiO2, P/F ratio ..

ELIGIBILITY:
Inclusion Criteria:

* All adult COVID-19 patients (>18 years) admitted to the ICU between 01/02/2020 and 31/07/2021 with a laboratory confirmation of COVID-19 infection with a positive result on polymerase chain reaction (PCR) assays of nasopharyngeal swab samples or bronchoalveolar lavage

Exclusion Criteria:

* All adult patients admitted for other reasons to the ICU (no COVID-19 pneumonia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult COVID-19 patients (>18 years) admitted to the ICU between 01/02/2020 and 31/07/2021 with a laboratory confirmation of COVID-19 infection with a positive result on polymerase chain reaction (PCR) assays of nasopharyngeal swab samples or bronchoalveolar lavage
Sampling Method: Non-Probability Sample
Enrollment: 295 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Mortality | through study completion, an average of 1 year
  mortality of patients during their stay at the ICU

SECONDARY OUTCOMES:
3 Months Mortality | 3 months after admission to ICU
  Mortality of patients
acute kidney injury | through study completion, an average of 1 year
  incidence of acute kidney injury
continous renal replacement therapy | through study completion, an average of 1 year
  incidence of continous renal replacement therapy
Length of stay in hospital | through study completion, an average of 1 year
  Length of stay in hospital
Length of stay in ICU | during ICU stay
  Length of stay in ICU

OTHER OUTCOMES:
Complications | through study completion, an average of 1 year
  description of possible complications after ECMO

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Madrid-Valero JJ, Ware J, Allen JM, Boughton CK, Hartnell S, Wilinska ME, Thankamony A, de Beaufort C, Schierloh U, Campbell FM, Sibayan J, Bocchino LE, Kollman C, Hovorka R, Gregory AM, Consortium K. Sleep Quality and Quantity in Caregivers of Children with Type 1 Diabetes Using Closed-Loop Insulin Delivery or a Sensor-Augmented Pump. Pediatr Diabetes. 2023 Jun 13;2023:7937007. doi: 10.1155/2023/7937007. eCollection 2023. PMID 40303271
- [Derived] Stessel B, Bin Saad M, Ullrick L, Geebelen L, Lehaen J, Timmermans PJ, Van Tornout M, Callebaut I, Vandenbrande J, Dubois J. Extracorporeal Membrane Oxygenation to Support COVID-19 Patients: A Propensity-Matched Cohort Study. Crit Care Res Pract. 2023 Jun 12;2023:5101456. doi: 10.1155/2023/5101456. eCollection 2023. PMID 37342313